CLINICAL TRIAL: NCT05020509
Title: Comparison of Intravascular Injection Rates During Cervical and Lumbar Medial Branch Block Using Touhy or Quincke Type Needle
Brief Title: Intravascular Injection Rates During Lumbar Medial Branch Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-07-014-001
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-08

CONDITIONS: Intravascular Injection
Keywords: intravascular injection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Touhy needle group (Active Comparator): medial branch block with touhy needle
  Interventions: Procedure: medial branch block
- Quincke needle group (Placebo Comparator): medial branch block with Quincke needle
  Interventions: Procedure: medial branch block

INTERVENTIONS:
Procedure: medial branch block — lumbar medial branch block
  Other Names: lumbar medial branch block

SUMMARY:
The purpose of this study is to compare using Toughy needle has an advantage of reducing the incidence of vasucular puncture during lumbar medial branch block.

DETAILED DESCRIPTION:
In previous reports, the use of Toughy needle was thought to reduce the incidence of intravascular injection during lumbar transforaminal injection. Blunt needles with a pencil point tip, such as Whitacre needles, are not as sharp at their tip as are Quincke needles, which have bevels. Toughy or blunt needles may therefore be less likely to penetrate a vessel during a procedure. Hence, the investigators postulated the incidence of intravenous uptake would be significantly lower using a Toughy needle than using a Quincke needle for lumbar medial branch block. To confirm the intravascular injection rates, the investigators used the real time fluoroscopy after injection of contrast medium.

The goal of this study was to compare the incidence of intravascular injection rate betweeen Toughy and Quincke needles using real time fluoroscopy during lumbar medial branch block

ELIGIBILITY:
Inclusion Criteria:

* facet joint arthropathy

Exclusion Criteria:

* allergy to local anesthetics or contrast medium
* pregnancy
* spine deformity
* neurologic abnormality

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
incidence of intravascular injection | 1 minute after finishing lumbar medial branch block
  incidence of intravascular injection during lumbar medial branch block

SECONDARY OUTCOMES:
time required to complete lumbar medial branch block | Baseline, 1 second after the completion of lumbar medial branch block
  time required to complete lumbar medial branch block
radiation amout to complete lumbar medial branch block | Baseline, 1 second after the completion of lumbar medial branch block
  radiation amout to complete lumbar medial branch block

CONTACTS AND LOCATIONS:
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No